CLINICAL TRIAL: NCT06668389
Title: Sodium-Glucose Cotransporter 2 Inhibitors for Repaired Tetralogy of Fallot Patients for Enhancement of Cardio-Pulmonary Status Trial (STEPS Trial)
Brief Title: Sodium-Glucose Cotransporter 2 Inhibitors for Repaired Tetralogy of Fallot Patients for Enhancement of Cardio-Pulmonary Status Trial
Acronym: STEPS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Chun Ka, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEPS; HKU / HA HKW IRB (Other: HKU / HA HKW IRB)
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Congenital Heart Disease; Repaired Tetralogy of Fallot (rTOF); Pulmonary Regurgitation; Sodium-glucose Cotransporter 2 (SGLT2) Inhibitor; Dapagliflozin (Forxiga)
Keywords: Congenital Heart Disease; Repaired Tetralogy of Fallot (rTOF); Pulmonary Regurgitation; Sodium-glucose cotransporter 2 (SGLT2) inhibitor; Dapagliflozin (Forxiga)
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Valve Insufficiency | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SGLT2 inhibitor Group (Experimental): Dapagliflozin 10mg once daily orally from Visit 1 (Week 1) to Visit 3 (Week 12 ± 1)
  Interventions: Drug: SGLT2 inhibitor (Dapagliflozin 10mg)
- Control Group (No Intervention): Routine care

INTERVENTIONS:
Drug: SGLT2 inhibitor (Dapagliflozin 10mg) — Subjects in SGLT2 inhibitor Group will take dapagliflozin 10mg once daily orally from Visit 1 (Week 1) to Visit 3 (Week 12 ± 1)
  Arms: SGLT2 inhibitor Group

SUMMARY:
Repaired Tetralogy of Fallot (rTOF) is the leading cause of congenital cyanotic heart disease worldwide, involving up to 7-10% of congenital heart disease. With advances in open-heart surgical repair techniques and medical therapies, there is a significant increase in patients with rTOF surviving till late adulthood. One sequalae that nearly all rTOF patients develop during their lifetime is significant pulmonary regurgitation. Pulmonary regurgitation causes progressive right ventricular dilatation and systolic dysfunction, which in turn impairs cardio-pulmonary function and overall survival.

There is currently no pharmacological therapy proven to improve cardio-pulmonary function in rTOF patients. In a double-blind, placebo controlled, randomized controlled trial involving 33 rTOF patients, the use of beta-adrenergic receptor blocker Bisoprolol failed to improve maximal oxygen uptake (VO2 max) in the treatment group. Furthermore, there was no significant change in dimension of right ventricle on cardiac imaging, or heart failure biomarkers including brain natriuretic peptide (BNP) and atrial natriuretic peptide (ANP). In the APPROPRIATE trial involving 64 patients, angiotensin-converting-enzyme inhibitor (ACEI) Ramipril similarly failed to improve VO2 max despite an improved right ventricular long-axis shortening. In REDEFINE trial, 95 rTOF patients were randomized in to receive angiotensin receptor blocker (ARB) Losartan and control. At the end of study, there was no significant difference between the two groups in VO2 max, right ventricular ejection fraction, and other key outcomes.

Sodium-glucose cotransporter 2 (SGLT2) inhibitor is a promising therapy for rTOF patients. Clinical trials consistently demonstrated that SGLT2 inhibitors reduce heart failure hospitalization and mortality among patients with heart failure with or without diabetes mellitus. There have been growing body of evidence that demonstrate that SGLT2 inhibitors improve right ventricular function. In a preclinical study of rat with pulmonary hypertension induced right ventricular failure, empagliflozin was found to reduce pulmonary pressure, alleviate right ventricular hypertrophy and reduce myocardial fibrosis. In a pilot study involving 10 patients with adult congenital heart disease and systemic right ventricular failure, SGLT2 inhibitors improved cardio-pulmonary function as reflected by 6-minute walk test performance and New York Heart Association functional status. Most recently, investigators from DAPA-SERVE randomized controlled trial reported that among 92 patients with systemic right ventricular failure, those randomized to receive SGLT2 inhibitors had superior systemic right ventricular function with larger fractional area change (FAC) and more negative free-wall global longitudinal strain. Nevertheless, as these trials involve patients with right ventricular connections to the systemic circulation rather than pulmonary circulation in rTOF, it is uncertain whether the trial results can be extrapolated to the rTOF population. The critical knowledge gap our proposed randomized controlled trial seeks to address is whether SGLT2 inhibitors improve cardio-pulmonary function in rTOF patients.

DETAILED DESCRIPTION:
Patients with repaired TOF fulfilling inclusion and exclusion criteria will be recruited from Queen Mary Hospital, Hong Kong.

Patients who fulfill the inclusion and exclusion criteria will be interviewed by research staff and given a detailed explanation of the clinical trial. Written informed consent will be obtained if the patient agrees to enroll in the trial.

Assessments will be performed at Visit 1 (week 1): Review of medical history and history taking, Physical examination of vital signs (including blood pressure, pulse rate, and oxygen saturation by pulse oximetry), and cardiovascular system (12-lead electrocardiography (ECG), Blood tests (if not already done within 3 months): Complete blood count, Renal function test, Liver function test, Calcium and phosphate levels, N-terminal pro b-type natriuretic peptide (Nt-pro-BNP), High sensitive troponin T, Creatinine kinase, Hemoglobin A1c (HbA1c), Fasting glucose, Lipid profile , Erythropoietin, Multi-omic studies including proteomics, metabolomics, and lipidomics, Genetic test and geneticist consultation, Echocardiography (if not already done within 3 years), Cardiopulmonary test (CPX), Urine pregnancy test in women of childbearing age.

Randomization will be performed on the day of recruitment. An allocation sequence will be generated prior to initiation of the clinical trial using random numbers generated by computer. After entering a subject's information on the clinical trial system, the allocated group for the subject will be revealed. If a subject found to be ineligible for the clinical trial after randomization, the original assignment will be allocated to the next eligible subject. Subjects will be randomized in a 1:1 ratio to 1 of the 2 treatment arms:

1. SGLT2 inhibitor Group: Dapagliflozin 10mg once daily orally from Visit 1 (Week 1) to Visit 3 (Week 12 ± 1)
2. Control Group: Routine care.

CPX will be performed on Visit 1 (week 4 ± 1) and Visit 3 (week 12 ± 1) under supervision of cardiologist blinded to randomization results. VO2 max, which represent the maximal amount of oxygen consumed during peak exercise, will be measured. In addition, other parameters including metabolic equivalents (METs) achieved, oxygen pulse, anaerobic threshold (VO2 AT), ventilatory equivalent for oxygen (VE/VO2) will be evaluated. Participant will concurrently be Apple Watch Series 9 (Apple, USA) smartwatch for pre- and post-SaO2 and VO2max assessment.

Echocardiography will be performed on Visit 1 and Visit 3 by independent echocardiographer blinded to randomization result. Right ventricular function will be assessed by measuring fractional area change (FAC), tricuspid annular plane systolic excursion (TAPSE), lateral tricuspid annulus peak systolic velocity (RVS'). Right ventricular diastolic diameter including basal (RVD1), mid ventricle (RVD2) and longitudinal (RVD3) will be measured. Tricuspid regurgitation severity will be graded using vena contracta with <0.2 cm as mild, 0.2-0.6 cm as moderate, and ≥0.7 cm as severe. Pulmonary regurgitation severity will be graded using semi-quantitative approach using right ventricular outflow view and parasternal short axis view with pressure half time <100 ms to be graded as severe.

ELIGIBILITY:
Inclusion Criteria:

* rTOF
* Aged 18 years or above
* Voluntarily agrees to participate in the clinical trial and provide written informed consent

Exclusion Criteria:

* Heart failure with reduced ejection fraction (HFrEF) with LVEF < 40%
* Planned cardiac and/or non-cardiac surgery in 3 months
* Chronic kidney disease stages 4 to 5
* Unable to perform cardiopulmonary test
* Recent use of SGLT2 inhibitors within 6 months
* Known hypersensitivity to SGLT2 inhibitors
* History of diabetic ketoacidosis
* Recent symptomatic hypoglycaemia within 6 months
* Insulin dependent diabetes mellitus
* History of perineum infection
* Recent urinary tract infection within 6 months
* Recent genital infection within 6 months
* Other known contraindication to SGLT2 inhibitor
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2 max) on cardiopulmonary exercise (CPX) at 3 months | At Visit 3 (3 months)
  Efficacy of SGLT2 inhibitors for improving cardiopulmonary function as assessed the maximal oxygen uptake (VO2 max) on cardiopulmonary exercise testing in rTOF patients at 3 months

SECONDARY OUTCOMES:
Right ventricular systolic function and dimension | At Visit 3 (3 months)
  Effect of SGLT2 inhibitors on right ventricular dimension and function in rTOF patients as assessed by performing echocardiography at 3 months
Pulmonary and tricuspid regurgitation severity | At Visit 3 (3 months)
  Effect of SGLT2 inhibitors on as pulmonary and tricuspid regurgitation severity as assessed by echocardiography at 3 months
Other cardiopulmonary test (CPX) parameters | At Visit 3 (3 months)
  Metabolic equivalents (METs) achieved, oxygen pulse, anaerobic threshold (VO2 AT), and ventilatory equivalent for oxygen (VE/VO2) are assessed during CPX for effect of of SGLT2 inhibitors in rTOF patients
Cardiac biomarkers level | At Visit 3 (3 months)
  Cardiac biomarkers level, including NT-proBNP and high sensitive troponin T in rTOF patients at 3 months as assessed via blood tests for effect of SGLT2 inhibitors
Minnesota Living with Heart Failure Questionnaire/ Kansa City Cardiomyopathy Questionnaire (KCCQ) score | At Visit 3 (3 months)
  Minnesota Living with Heart Failure Questionnaire/ Kansa City Cardiomyopathy Questionnaire (KCCQ) score as completed with rTOF patients for effect of SGLT2 inhibitors
Time to first occurrence of clinical events | At Visit 3 (3 months)
  Time to first occurrence of clinical events, including heart failure hospitalization, incident arrhythmia, and cardiovascular mortality in 3 months safety as assessed for tolerability of SGLT2 inhibitors in rTOF patients
Occurrence of adverse events | At Visit 3 (3 months)
  Occurrence of adverse events in 3 months as assessed for safety and tolerability SGLT2 inhibitors in rTOF patients

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ka Dr Wong, Clinical Assistant Professor, Principal Investigator — The University of Hong Kong/ Department of Medicine, Queen Mary Hospital
Locations (1):
- Department of Medicine, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gong Z, Xing D, Wu R, Zhang S, Ye C, Chen Y, Liu X, Chen L, Wang T. Prognostic value of N-terminal pro-form B-type natriuretic peptide (NT-proBNP) in patients with congenital heart disease undergoing cardiac surgery: a systematic review and meta-analysis of cohort studies. Cardiovasc Diagn Ther. 2022 Dec;12(6):853-867. doi: 10.21037/cdt-22-155. PMID 36605072
- [Background] Wadey CA, Weston ME, Dorobantu DM, Pieles GE, Stuart G, Barker AR, Taylor RS, Williams CA. The role of cardiopulmonary exercise testing in predicting mortality and morbidity in people with congenital heart disease: a systematic review and meta-analysis. Eur J Prev Cardiol. 2022 Mar 25;29(3):513-533. doi: 10.1093/eurjpc/zwab125. PMID 34405863
- [Background] Neijenhuis RML, Nederend M, Jongbloed MRM, Kies P, Rotmans JI, Vliegen HW, Jukema JW, Egorova AD. The potential of sodium-glucose cotransporter 2 inhibitors for the treatment of systemic right ventricular failure in adults with congenital heart disease. Front Cardiovasc Med. 2023 Jun 26;10:1093201. doi: 10.3389/fcvm.2023.1093201. eCollection 2023. PMID 37435053
- [Background] Fusco F, Scognamiglio G, Abbate M, Merola A, Grimaldi N, Ciriello GD, Sarubbi B. Dapagliflozin in Patients With a Failing Systemic Right Ventricle: Results From the DAPA-SERVE Trial. JACC Heart Fail. 2024 Apr;12(4):789-791. doi: 10.1016/j.jchf.2024.01.006. Epub 2024 Feb 28. No abstract available. PMID 38430085
- [Background] Wu J, Liu T, Shi S, Fan Z, Hiram R, Xiong F, Cui B, Su X, Chang R, Zhang W, Yan M, Tang Y, Huang H, Wu G, Huang C. Dapagliflozin reduces the vulnerability of rats with pulmonary arterial hypertension-induced right heart failure to ventricular arrhythmia by restoring calcium handling. Cardiovasc Diabetol. 2022 Sep 28;21(1):197. doi: 10.1186/s12933-022-01614-5. PMID 36171554
- [Background] Axelsen JS, Nielsen-Kudsk AH, Schwab J, Ringgaard S, Nielsen-Kudsk JE, de Man FS, Andersen A, Andersen S. Effects of empagliflozin on right ventricular adaptation to pressure overload. Front Cardiovasc Med. 2023 Dec 14;10:1302265. doi: 10.3389/fcvm.2023.1302265. eCollection 2023. PMID 38162132
- [Background] van den Bosch E, van Genuchten WJ, Luijnenburg SE, Duppen N, Kamphuis VP, Roos-Hesselink JW, Bartelds B, Roest AAW, Breur JMPJ, Blom NA, Boersma E, Koopman LP, Helbing WA. Associations between blood biomarkers, cardiac function and adverse outcome in a young tetralogy of Fallot cohort. Int J Cardiol. 2022 Aug 15;361:31-37. doi: 10.1016/j.ijcard.2022.04.065. Epub 2022 Apr 26. PMID 35487320
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2023 Oct 1;44(37):3627-3639. doi: 10.1093/eurheartj/ehad195. No abstract available. PMID 37622666
- [Background] Nunez J, Palau P, Dominguez E, Mollar A, Nunez E, Ramon JM, Minana G, Santas E, Facila L, Gorriz JL, Sanchis J, Bayes-Genis A. Early effects of empagliflozin on exercise tolerance in patients with heart failure: A pilot study. Clin Cardiol. 2018 Apr;41(4):476-480. doi: 10.1002/clc.22899. Epub 2018 Apr 17. PMID 29663436
- [Background] Chen K, Nie Z, Shi R, Yu D, Wang Q, Shao F, Wu G, Wu Z, Chen T, Li C. Time to Benefit of Sodium-Glucose Cotransporter-2 Inhibitors Among Patients With Heart Failure. JAMA Netw Open. 2023 Aug 1;6(8):e2330754. doi: 10.1001/jamanetworkopen.2023.30754. PMID 37615988
- [Background] Santos-Gallego CG, Vargas-Delgado AP, Requena-Ibanez JA, Garcia-Ropero A, Mancini D, Pinney S, Macaluso F, Sartori S, Roque M, Sabatel-Perez F, Rodriguez-Cordero A, Zafar MU, Fergus I, Atallah-Lajam F, Contreras JP, Varley C, Moreno PR, Abascal VM, Lala A, Tamler R, Sanz J, Fuster V, Badimon JJ; EMPA-TROPISM (ATRU-4) Investigators. Randomized Trial of Empagliflozin in Nondiabetic Patients With Heart Failure and Reduced Ejection Fraction. J Am Coll Cardiol. 2021 Jan 26;77(3):243-255. doi: 10.1016/j.jacc.2020.11.008. Epub 2020 Nov 13. PMID 33197559
- [Background] Chowdhury B, Luu AZ, Luu VZ, Kabir MG, Pan Y, Teoh H, Quan A, Sabongui S, Al-Omran M, Bhatt DL, Mazer CD, Connelly KA, Verma S, Hess DA. The SGLT2 inhibitor empagliflozin reduces mortality and prevents progression in experimental pulmonary hypertension. Biochem Biophys Res Commun. 2020 Mar 26;524(1):50-56. doi: 10.1016/j.bbrc.2020.01.015. Epub 2020 Jan 21. PMID 31980166
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Bokma JP, Winter MM, van Dijk AP, Vliegen HW, van Melle JP, Meijboom FJ, Post MC, Berbee JK, Boekholdt SM, Groenink M, Zwinderman AH, Mulder BJM, Bouma BJ. Effect of Losartan on Right Ventricular Dysfunction: Results From the Double-Blind, Randomized REDEFINE Trial (Right Ventricular Dysfunction in Tetralogy of Fallot: Inhibition of the Renin-Angiotensin-Aldosterone System) in Adults With Repaired Tetralogy of Fallot. Circulation. 2018 Apr 3;137(14):1463-1471. doi: 10.1161/CIRCULATIONAHA.117.031438. Epub 2017 Dec 8. PMID 29222139
- [Background] Babu-Narayan SV, Uebing A, Davlouros PA, Kemp M, Davidson S, Dimopoulos K, Bayne S, Pennell DJ, Gibson DG, Flather M, Kilner PJ, Li W, Gatzoulis MA. Randomised trial of ramipril in repaired tetralogy of Fallot and pulmonary regurgitation: the APPROPRIATE study (Ace inhibitors for Potential PRevention Of the deleterious effects of Pulmonary Regurgitation In Adults with repaired TEtralogy of Fallot). Int J Cardiol. 2012 Feb 9;154(3):299-305. doi: 10.1016/j.ijcard.2010.09.057. Epub 2010 Oct 22. PMID 20970202
- [Background] Norozi K, Bahlmann J, Raab B, Alpers V, Arnhold JO, Kuehne T, Klimes K, Zoege M, Geyer S, Wessel A, Buchhorn R. A prospective, randomized, double-blind, placebo controlled trial of beta-blockade in patients who have undergone surgical correction of tetralogy of Fallot. Cardiol Young. 2007 Aug;17(4):372-9. doi: 10.1017/S1047951107000844. Epub 2007 Jun 18. PMID 17572925
- [Background] Muller J, Hager A, Diller GP, Derrick G, Buys R, Dubowy KO, Takken T, Orwat S, Inuzuka R, Vanhees L, Gatzoulis M, Giardini A. Peak oxygen uptake, ventilatory efficiency and QRS-duration predict event free survival in patients late after surgical repair of tetralogy of Fallot. Int J Cardiol. 2015 Oct 1;196:158-64. doi: 10.1016/j.ijcard.2015.05.174. Epub 2015 Jun 2. PMID 26114442
- [Background] Ghonim S, Gatzoulis MA, Ernst S, Li W, Moon JC, Smith GC, Heng EL, Keegan J, Ho SY, McCarthy KP, Shore DF, Uebing A, Kempny A, Alpendurada F, Diller GP, Dimopoulos K, Pennell DJ, Babu-Narayan SV. Predicting Survival in Repaired Tetralogy of Fallot: A Lesion-Specific and Personalized Approach. JACC Cardiovasc Imaging. 2022 Feb;15(2):257-268. doi: 10.1016/j.jcmg.2021.07.026. Epub 2021 Oct 13. PMID 34656466
- [Background] Forman J, Beech R, Slugantz L, Donnellan A. A Review of Tetralogy of Fallot and Postoperative Management. Crit Care Nurs Clin North Am. 2019 Sep;31(3):315-328. doi: 10.1016/j.cnc.2019.05.003. Epub 2019 Jul 5. PMID 31351553